CLINICAL TRIAL: NCT07063316
Title: Effect of SGLT2 Inhibitors on Renal Anemia and Its Management in Patients With CKD in Japan
Brief Title: SGLT2 Inhibitors and Renal Anemia in Japan: RWD
Status: Active, not recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0387
Record Dates: First submitted 2025-06-24; First posted 2025-07-14 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SGLT2 inhibitor users
  Interventions: Drug: SGLT2 inhibitor
- SGLT2 inhibitor non-users

INTERVENTIONS:
Drug: SGLT2 inhibitor — SGLT2 inhibitor
  Groups: SGLT2 inhibitor users

SUMMARY:
The objectives of the study are:

1. To compare the risk and timing of anemia onset between Sodium-Glucose Co-Transporter-2 (SGLT2) inhibitor users and non-users in patients with chronic kidney disease (CKD) from the index date to first event occurrence or the end date of each individual's follow-up.
2. To compare the following outcomes from the index date to 731 days (24 months) or the end date of each individual's follow-up:

A) Longitudinal changes in laboratory values between SGLT2 inhibitor users and non-users in patients with CKD.

B) Prescription patterns and treatment regimens for anemia between SGLT2 inhibitor users and non-users in patients with CKD, including analysis of medication types, dosing strategies, and duration of treatments.

C) Anemia-related healthcare costs between SGLT2 inhibitor users and non-users.

ELIGIBILITY:
Inclusion Criteria:

1. Have two consecutive estimated glomerular filtration rate (eGFR) measurements < 60 mL/min/1.73 m2 at least 92 days apart between October 1, 2013 and October 31, 2022.
2. Aged 18 years or older at the index date.

Exclusion Criteria:

1. Have less than 183 days of record history before the index date.
2. Have a any prescription record for an SGLT2 inhibitor at the index date or within 183 days before the index date
3. Have evidence of anemia at the index date or within 183 days before the index date.

   * Hemoglobin (Hb) < 13.0 g/dL for men or < 12.0 g/dL for women
   * Hematocrit (Ht) < 39% for men or < 36% for women
   * Have a history of prescribed anemia-related medications and treatments at the index date or within 183 days before the index date.
4. Have evidence of anemia-causing conditions other than chronic kidney disease (CKD) at the index date or within 183 days before the index date.
5. Confirm at least one instance of hemodialysis, peritoneal dialysis, or kidney transplantation at the index date or within 183 days before the index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic kidney disease patients registered in the Medical Data Vision (MDV) database in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to the first occurrence of anemia (composite anemia outcomes) | From the index date to first event occurrence or the end date of each individual's follow-up, up to 13 years
  The composite of anemia outcomes is defined as any of the following:
  * Hb < 13.0 g/dL for men or < 12.0 g/dL for women
  * Clinical diagnosis of anemia using ICD-10 diagnosis codes
  * Initiation of anemia treatment (Erythropoiesis-Stimulating Agents (ESAs), Hypoxia-Inducible Factor-Prolyl Hydroxylase (HIF-PH) inhibitors, iron preparations, or red blood cell (RBC) transfusion

SECONDARY OUTCOMES:
Number of administered doses of ESA, HIF-PH inhibitors, iron preparations, and RBC transfusions | Up to 24 months
  Erythropoiesis-Stimulating Agents (ESAs) Hypoxia-Inducible Factor-Prolyl Hydroxylase (HIF-PH) Red blood cell (RBC) transfusions
Anemia-related healthcare costs | Up to 24 months
  Anemia-related medical costs are defined as the sum of direct medical costs associated with the treatment of anemia. These costs will include medication costs and costs related to RBC transfusion.
Frequency of administration of ESA, HIF-PH inhibitors, iron preparations, and RBC transfusions | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Boehringer Ingelheim Co ., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com